CLINICAL TRIAL: NCT05737797
Title: Non-Invasive Diagnosis of Endometrial Cancer
Acronym: NIECE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP221027
Record Dates: First submitted 2022-12-26; First posted 2023-02-21 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Next-generation sequencing; Screening; Microsatellite instability
MeSH Terms: conditions — Endometrial Neoplasms; Microsatellite Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endometrial cancer patients (Experimental): Endometrial cancer patients Cervical cytology during surgical intervention.
  Interventions: Procedure: cervical cytology during surgery.

INTERVENTIONS:
Procedure: cervical cytology during surgery. — Cervical cytology will be performed by the surgeon in the operating theatre before hysterectomy.

SUMMARY:
The study aims to determine whether next generation sequencing and microsatellite analysis of cervical cytology is sensitive for the detection of endometrial carcinoma.

DETAILED DESCRIPTION:
Definitive diagnosis of endometrial cancer relies on endometrial biopsy, in addition to imaging. Biopsy is however invasive and often painful, and its sensitivity in only moderate. Cervical cytology could be an alternative. This is a proof-of-concept study. The investigators will carry out next generation sequencing of cervical cytology in patients with confirmed endometrial carcinoma, in order to determine whether activating variants are identified. About 15% of endometrial carcinomas are microsatellite instable (MSI). The investigators will therefore also carry out MSI analysis using MSICare in the subset of cases with MMR-deficient cancer.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial cancer requiring hysterectomy
* Patient covered by French social Security
* Patient capable of giving written informed consent

Exclusion Criteria:

- Chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Activating variants and MSI via cytology | 16 months
  proportion of cases in whom genetic activating variants and microsatellite instability are detected by cytology

SECONDARY OUTCOMES:
Type of variants | 16 months
  Variant details
Number of variants | 16 months
  Variant details
Frequency of variants | 16 months
  Variant details
Comparison with the proportion of variants seen on the pathological | 16 months
  Tumoral correlation
Comparison with the proportion of microsatellite instability detected on the pathological specimen. | 16 months
  Tumoral correlation

CONTACTS AND LOCATIONS:
Locations (1):
- Medical genetics department, Paris, France

IPD SHARING:
Plan to Share IPD: No